CLINICAL TRIAL: NCT04373187
Title: A Phase 1, Randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Two Different Dose Concentrations of CC-93538 in Healthy Adult Subjects
Brief Title: Study to Evaluate the Pharmacokinetic Comparability of CC-93538 From Two Different Drug Concentrations in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC-93538-CP-002; U1111-1250-3915 (Other: WHO)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers
Keywords: CC-93538; Healthy Subjects; PK comparability between two different dose concentrations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CC-93538, 180mg/mL (Experimental): 26 healthy subjects will receive one injection of 2mL, 180mg/mL CC-93538
  Interventions: Drug: CC-93538
- CC-93538, 150mg/mL (Experimental): 26 healthy subjects will receive 2 injections of 1.2mL, 150mg/mL CC-93538
  Interventions: Drug: CC-93538

INTERVENTIONS:
Drug: CC-93538 — one injection of 2mL
Drug: CC-93538 — two injections of 1.2mL
  Arms: CC-93538, 150mg/mL

SUMMARY:
This is an open-label, randomized, parallel design study to evaluate the PK comparability, safety, tolerability and immunogenicity of a single SC dose of 360 mg CC 93538 using two different drug concentrations, 180 mg/mL and 150 mg/mL, in healthy adult subjects.

A total of approximately 52 subjects will be enrolled and randomized 1:1 to receive a single 360 mg SC dose of CC-93538 using either 180 mg/mL (1 injection of 2 mL) or 150 mg/mL (2 injections of 1.2 mL each) drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must be male or non-pregnant female, aged ≥ 18 and ≤ 55 years of age at the time of signing the ICF.
2. Subject must have a body weight of at least 40 kg; a BMI ≥ 18 and ≤ 30 kg/m2 at screening and Day -1.
3. Subject must be in good health, as determined by the Investigator on the basis of medical history, clinical laboratory safety test results, vital signs, 12-lead ECG, and PE at Screening.
4. Female subjects not of childbearing potential must:

   1. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or
   2. Postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle stimulating hormone [FSH] level in the postmenopausal range according to the laboratory used at Screening); FSH to be performed at the discretion of the Investigator in consultation with the Medical Monitor.

   Females of child-bearing potential (FCBP) must agree to practice a highly effective method of contraception throughout the study and for 5 months after the last dose of investigational product (IP). FCBP is a female who 1) has achieved menarche at some point; 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

   Acceptable methods of birth control in this study are the following:
   * Combined hormonal (containing oestrogen and progestogen) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable or implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomised partner
   * Sexual abstinence
5. Subjects must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted, and must be able to comply with the requirements of the study, including the study visit schedule and other protocol requirements. Must be able to communicate with the Investigator and to understand and adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical history/condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition (acute or chronic) including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, ifkn own (whichever was longer).
5. Subject has previously received CC-93538 treatment (formerly known as RPC4046 and ABT-308).
6. Subject has a history of infection within 30 days of dosing on Day 1.
7. Subject has a history of drug or alcohol abuse (as defined by the investigator), or addiction within 6 months prior to Screening.
8. Subject has a positive urine drug test, or positive alcohol urine or breath test at Screening or on Day -1.
9. Subject has donated greater than 400 mL of blood within 60 days prior to Day 1.
10. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
11. Subject has a history of clinically significant allergic reaction to any drug, biologic, food, or vaccine.
12. Subject has a history of major immunologic reaction (such as anaphylactic reaction, anaphylactoid reaction, or serum sickness) to any IgG-containing agent.
13. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to dosing (Day 1) and throughout the study
14. Subject has tattoos (> 25% of their body) or other skin markings (eg, scars) that, in the opinion of the investigator, would prevent visualization of dermatologic changes due to study treatment
15. Subject has an active parasitic/helminthic infection or suspected parasitic helminthic infection. Subjects with suspected infections may participate if clinical and laboratory
16. Subject has been diagnosed with or is being treated for a clinical schistosomiasis.
17. Subject has a history of tuberculosis, or listeriosis.
18. Subject has a history of hereditary fructose intolerance.
19. Subject is, for any reason, deemed by the Investigator to be inappropriate for this study.
20. Subject has received any drug by injection within 30 days of Day 1.
21. Subject has poor peripheral venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - AUC0-∞ | From Day 0 to Day 105
  Area under the concentration-time curve calculated from time zero to infinity
Pharmacokinetic - Cmax | From Day 0 to Day 105
  Maximum observed concentration of drug

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment to Day 105
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Pharmacokinetic - AUC0-last | From Day 0 to Day 105
  Area under the concentration-time curve calculated from time zero to the last measured time point
Pharmacokinetic - tmax | From Day 0 to Day 105
  Time to Cmax
Pharmacokinetic - t½ | From Day 0 to Day 105
  Terminal elimination half-life
Pharmacokinetic - CL/F | From Day 0 to Day 105
  Apparent clearance of drug from serum after extravascular administration
Pharmacokinetic - Vz/F | From Day 0 to Day 105
  Apparent volume of distribution during the terminal phase

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/